CLINICAL TRIAL: NCT02748538
Title: A Randomised Controlled Trial to Evaluate the Effect of Face-down Posturing on Retinal Displacement and Distortion Following Retinal Detachment Repair
Brief Title: The Posturing After Retinal Detachment (Post RD) Trial
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CHAD1032
Record Dates: First submitted 2016-03-30; First posted 2016-04-22 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2016-03

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Face Down: To posture in the face down position for the first 24 hours following surgery.
- Position to Support the Break: The head is positioned so that the retinal breaks (which caused the retinal detachment) are positioned at the highest point of the eye and well supported by the intra-ocular gas bubble left within the eye at the completion of surgery.

SUMMARY:
A randomised controlled trial to evaluate the effect of face-down posturing on retinal displacement and distortion following retinal detachment repair.

DETAILED DESCRIPTION:
During the surgical repair of a retina detachment, a gas bubble is inserted into the eye to keep the retina flat. Following this, it is common to ask patients to adopt a certain head position for a set period of time after their operation. This is known as posturing. It is thought that by adopting a certain head position/posturing, the bubble aids re-attachment of the retina. However, when the retinal detachment involves the macula (central portion of the retina) it has been shown that the retina can shift (or displace) post-operatively, leading to distortion in the patient's vision.

The purpose of this study is to investigate whether adopting different head positions following surgery for macula involving retinal detachments, can reduce retinal displacement and visual distortion. The investigators plan to recruit 368 patients. Patients will be in follow up for a period of six months. The study will be operational at two different hospitals in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Fovea-involving rhegmatogenous retinal detachment
* History of central visual loss within the past 14 days
* Patients undergoing vitrectomy and gas surgery, under local anaesthetic
* Able to give informed consent
* 18 years old and over

Exclusion Criteria:

* Previous vitrectomy or cryo-buckle surgery
* Retinal detachment surgery requiring silicone oil tamponade
* Existing ophthalmic condition which limits the patient's visual acuity (BCVA 6/36 or worse)
* Inability to posture post-operatively or commit to follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with macula-involving rhegmatogenous retinal detachment
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
To assess the proportion of patients in each treatment group with retinal displacement at 26 weeks after surgery | 26 Weeks
  The proportion of patients in each treatment group with retinal displacement at 26 weeks after surgery

SECONDARY OUTCOMES:
To assess the degree of retinal displacement on autofluorescence imaging | 26 Weeks
  Degree of retinal displacement on autofluorescence imaging at 26 weeks
To assess proportion of patients in each group with retinal displacement at 8 weeks | Eight weeks
  The proportion of patients in each group with retinal displacement at 8 weeks after surgery.
To report the mean (SD)/median (IQR) ETDRS visual acuity score at two different time-points | Eight and 26 weeks
  To report the mean (SD)/median (IQR) ETDRS visual acuity score at 8 and 26 weeks after surgery in each treatment group
To report the mean(SD)/median(IQR) Objective distortion score at two different time-points | Eight and 26 weeks
  To report the mean(SD)/median(IQR) Objective distortion score at 8 and 26 weeks after surgery in each treatment group - with Objective distortion measured with D Charts
To report the mean (SD) / median (IQR) Visual function score as measured using the Visual Function Questionnaire | 26 Weeks
  To report the mean (SD) / median (IQR) Visual function score as measured using the Visual Function Questionnaire (NEI Visual Function Questionnaire 25) in each treatment group at 26 weeks after surgery.

OTHER OUTCOMES:
To assess subjective distortion by comparing patient's scores from the distortion questionnaire | Eight and 26 weeks
  Subjective distortion: a comparison of patient's scores in the distortion questionnaire at 8 & 26 weeks.
To assess the persistence of post-operative distortion: paired comparisons of subjective & objective distortion at two separate time-points | Eight and 26 weeks
  Persistence of post-operative distortion: paired comparisons of subjective & objective distortion at 8 and 26 weeks.
To assess the correlation between retinal displacement and distortion | Eight or 26 weeks
  Correlation between retinal displacement and distortion: the correlation between the incidence retinal displacement on autofluorescence imaging and distortion (questionnaire and D chart assessments) at 8 or 26 weeks.
To assess the relationship of exploratory outcome parameters at 26 weeks to self-recorded posturing diary | 26 Weeks
  Relationship of exploratory outcome parameters at 26 weeks to self-recorded posturing diary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casswell EJ, Yorston D, Lee E, Heeren TFC, Harris N, Zvobgo TM, Tarafdar S, Xing W, Bourmpaki E, Bunce C, Keane P, Charteris DG. Effect of Face-Down Positioning vs Support-the-Break Positioning After Macula-Involving Retinal Detachment Repair: The PostRD Randomized Clinical Trial. JAMA Ophthalmol. 2020 Jun 1;138(6):634-642. doi: 10.1001/jamaophthalmol.2020.0997. PMID 32297923